CLINICAL TRIAL: NCT02522676
Title: Comparison of Success Rates, Complication Rates and Injury to Kidneys of Conventional PCNL, Mini PCNL, Ultra-mini PCNL, Micro PCNL, RIRS and ESWL in the Treatment of Lower Pole and Renal Pelvis Stone(s)
Brief Title: Evaluation of Different Treatment Modalities for Lower Pole and Renal Pelvis Stones
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to surgeons' unwillingness to randomize patients into different treatments
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Murat AKAND, Assistant Professor, M.D., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-PCNL-LPRPS-01
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Kidney Stones
Keywords: kidney stone; percutaneous nephrolithotripsy; retrograde intrarenal surgery; extracorporeal shock wave lithotripsy; mini PCNL; ultra-mini PCNL; micro PCNL
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Conventional PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo conventional percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Mini PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo mini percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Ultra-mini PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo ultra-mini percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Micro PCNL (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo micro percutaneous nephrolithotripsy.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Retrograde intrarenal surgery (Active Comparator): Endoscopic kidney stone surgery: Patients will undergo retrograde intrarenal surgery.
  Interventions: Procedure: Endoscopic kidney stone surgery
- Extracorporeal shock wave lithotripsy (Active Comparator): Non-invasive kidney stone treatment: Patients will undergo extracorporeal shock wave lithotripsy.
  Interventions: Procedure: Non-invasive kidney stone treatment

INTERVENTIONS:
Procedure: Endoscopic kidney stone surgery — Conventional PCNL will be performed.
  Arms: Conventional PCNL
Procedure: Endoscopic kidney stone surgery — Mini PCNL will be performed.
  Arms: Mini PCNL
Procedure: Endoscopic kidney stone surgery — Ultra-mini PCNL will be performed.
  Arms: Ultra-mini PCNL
Procedure: Endoscopic kidney stone surgery — Micro PCNL will be performed.
  Arms: Micro PCNL
Procedure: Endoscopic kidney stone surgery — Retrograde intrarenal surgery will be performed.
  Arms: Retrograde intrarenal surgery
Procedure: Non-invasive kidney stone treatment — Extracorporeal shock wave will be performed.
  Arms: Extracorporeal shock wave lithotripsy

SUMMARY:
It is aimed to evaluate the treatment results, rates of success and complications, and injury given to the kidney by measuring preoperative and postoperative blood urea, creatinine, Cystatin C and Netrin-1 levels and urine Cystatin C and Netrin-1 levels in patients with lower pole or renal pelvis stone(s) undergoing either one of the treatment modalities including conventional percutaneous nephrolithotripsy (PCNL), mini PCNL, ultra-mini PCNL, micro PCNL, retrograde intrarenal surgery (RIRS) and extracorporeal shock wave lithotripsy (ESWL).

DETAILED DESCRIPTION:
In this study, the demographic and preoperative data, imaging data, operative data and postoperative follow-up data will be prospectively recorded according to the patient information forms for the patients with lower pole and/or renal pelvis stone(s) who will undergo either one of the treatment modalities including conventional PCNL, mini PCNL, ultra-mini PCNL, micro PCNL, RIRS and ESWL.

A total of 300 (three hundred) patients, aging between 18 and 70 years, with similar stone size and location are being planned to be enrolled into the study; and will be prospectively randomized into one of six groups with a 1:1 ratio. By this means, conventional PCNL will performed to 50 (fifty) patients, mini PCNL will be performed to 50 (fifty) patients, ultra-mini PCNL will be performed to 50 (fifty) patients, micro PCNL will be performed to 50 (fifty) patients, while 50 (fifty) patients will undergo RIRS and 50 (fifty) patients will undergo ESWL.

Preoperatively, blood Cystatin C and Netrin-1, and urine Neutrophil gelatinase-associated lipocalin (NGAL), Cystatin C and Netrin-1 levels will be measured. After the treatments, blood Cystatin C and Netrin-1 levels at postoperative 6th, 12th, 24th and 48th hours will be recorded. Cystatin C and Netrin-1 levels in urine will be measured at postoperative 12th and 24th hours, while urine NGAL levels will be measured at postoperative 12th and 72nd hours. Besides these, classical kidney function tests, namely blood urea and creatinine levels, will be measured preoperatively and postoperatively at 24th and 48th hours.

Parameters listed below will be also recorded and evaluated:

1. Preoperative general evaluation data: Age, height, weight, body-mass index, concomitant comorbidities, prescriptions used, history of operation(s), American Society of Anesthesiologists (ASA) score
2. Preoperative urological evaluation data: History of ESWL/PCNL/ureterorenoscopy (URS)/RIRS/open surgery, whole blood count, kidney function tests, automatic urine test, urine culture, preoperative imaging modality (KUB, US, CT), number-dimensions-localization-composition of stone(s), existence of hydronephrosis
3. Operative data: Access fluoroscopy duration, total access duration, total fluoroscopy duration, operation duration, use of double-J stent, preoperative complications
4. Number of previous ESWL seance, total duration of ESWL, number of shots during ESWL (if any)
5. Follow-up data: Urethral catheterization time, hospitalization time, need of any other treatment for being stone-free, time to full stone-free, duration to removal of double-J stent, existence of residual stone(s), formation of new stone(s), complications in late time, medical prophylaxis
6. Stone analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to undergo either conventional PCNL, mini PCNL, ultra-mini PCNL, micro PCNL, RIRS or ESWL due to kidney stone(s)
* Patients between 18 and 70 years old

Exclusion Criteria:

* Patients with unregulated diabetes mellitus and diabetic nephropathy
* Patients with a blood pressure higher than 140/80 mmHg despite use of antihypertensive drug(s) regularly
* Patients with chronic renal failure who need dialysis
* Patients who had prerenal, renal or postrenal acute kidney failure during the last 6 months
* Patients who had acute pyelonephritis during the last 6 months
* Patients younger than 18 years old or older than 70 years old
* Patients who had kidney surgery during the last 3 months and who have abnormal kidney functions
* Patients with ureteral stone who are planned to undergo endoscopic stone treatment at the same time
* Patients with a history of corticosteroid use during enrollment into the study or previous 3 months
* Patients with uncontrolled thyroid disease
* Patients who have a disease with rapid cell turn-over (like leukemia, lymphoma, etc.)
* Patients in whom PCNL/RIRS/ESWL cannot be performed due to any reason and the procedure is terminated
* Patients who are converted to open surgery due to any reason
* Patients with missing data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | Within the first 30 days after surgery/procedure
  Determination of any residual stone in the collecting system by using one of imaging modalities.

SECONDARY OUTCOMES:
Complication rate | Within the first 30 days after surgery/procedure
  Determination of any complications related to the surgery/procedure.
Blood Cystatin C level (mg/L) | Within the first 48 hours after surgery/procedure
  Determination of any impairment in renal function after the surgery/procedure by measuring blood Cystatin C level.
Blood Netrin-1 level (pg/mL) | Within the first 48 hours after surgery/procedure
  Determination of any impairment in renal function after the surgery/procedure by measuring blood Netrin-1 level.
Urine NGAL level (ng/mL) | Within the first 72 hours after surgery/procedure
  Determination of any impairment in renal function after the surgery/procedure by measuring urine NGAL level.
Urine Cystatin C level (mg/L) | Within the first 24 hours after surgery/procedure
  Determination of any impairment in renal function after the surgery/procedure by measuring urine Cystatin C level.
Urine Netrin-1 level (pg/mL) | Within the first 24 hours after surgery/procedure
  Determination of any impairment in renal function after the surgery/procedure by measuring urine Netrin-1 level.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Akand, M.D., Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skolarikos A, Straub M, Knoll T, Sarica K, Seitz C, Petrik A, Turk C. Metabolic evaluation and recurrence prevention for urinary stone patients: EAU guidelines. Eur Urol. 2015 Apr;67(4):750-63. doi: 10.1016/j.eururo.2014.10.029. Epub 2014 Nov 20. PMID 25454613
- [Background] de la Rosette J, Assimos D, Desai M, Gutierrez J, Lingeman J, Scarpa R, Tefekli A; CROES PCNL Study Group. The Clinical Research Office of the Endourological Society Percutaneous Nephrolithotomy Global Study: indications, complications, and outcomes in 5803 patients. J Endourol. 2011 Jan;25(1):11-7. doi: 10.1089/end.2010.0424. PMID 21247286
- [Background] Kamphuis GM, Baard J, Westendarp M, de la Rosette JJ. Lessons learned from the CROES percutaneous nephrolithotomy global study. World J Urol. 2015 Feb;33(2):223-33. doi: 10.1007/s00345-014-1367-5. Epub 2014 Aug 7. PMID 25100624
- [Background] Bader MJ, Gratzke C, Seitz M, Sharma R, Stief CG, Desai M. The "all-seeing needle": initial results of an optical puncture system confirming access in percutaneous nephrolithotomy. Eur Urol. 2011 Jun;59(6):1054-9. doi: 10.1016/j.eururo.2011.03.026. Epub 2011 Apr 1. PMID 21477921
- [Background] Desai MR, Sharma R, Mishra S, Sabnis RB, Stief C, Bader M. Single-step percutaneous nephrolithotomy (microperc): the initial clinical report. J Urol. 2011 Jul;186(1):140-5. doi: 10.1016/j.juro.2011.03.029. Epub 2011 May 14. PMID 21575966
- [Background] Hatipoglu NK, Tepeler A, Buldu I, Atis G, Bodakci MN, Sancaktutar AA, Silay MS, Daggulli M, Istanbulluoglu MO, Karatag T, Gurbuz C, Armagan A, Caskurlu T. Initial experience of micro-percutaneous nephrolithotomy in the treatment of renal calculi in 140 renal units. Urolithiasis. 2014 Apr;42(2):159-64. doi: 10.1007/s00240-013-0631-2. Epub 2013 Dec 13. PMID 24337646
- [Background] Desai J, Solanki R. Ultra-mini percutaneous nephrolithotomy (UMP): one more armamentarium. BJU Int. 2013 Nov;112(7):1046-9. doi: 10.1111/bju.12193. Epub 2013 Jul 11. PMID 23841665
- [Background] Resorlu B, Unsal A, Gulec H, Oztuna D. A new scoring system for predicting stone-free rate after retrograde intrarenal surgery: the "resorlu-unsal stone score". Urology. 2012 Sep;80(3):512-8. doi: 10.1016/j.urology.2012.02.072. Epub 2012 Jul 26. PMID 22840867
- [Background] Cepeda M, Amon JH, Mainez JA, Rodriguez V, Alonso D, Martinez-Sagarra JM. Flexible ureteroscopy for renal stones. Actas Urol Esp. 2014 Nov;38(9):571-5. doi: 10.1016/j.acuro.2014.03.014. Epub 2014 Jun 2. English, Spanish. PMID 24881777
- [Background] Gao X, Peng Y, Shi X, Li L, Zhou T, Xu B, Sun Y. Safety and efficacy of retrograde intrarenal surgery for renal stones in patients with a solitary kidney: a single-center experience. J Endourol. 2014 Nov;28(11):1290-4. doi: 10.1089/end.2014.0295. Epub 2014 Aug 6. PMID 24892920
- [Background] Palmero JL, Miralles J, Garau C, Nuno de la Rosa I, Amoros A, Benedicto A. Retrograde intrarenal surgery (RIRS) in the treatment of calyceal diverticulum with lithiasis. Arch Esp Urol. 2014 May;67(4):331-6. English, Spanish. PMID 24892394
- [Background] Aboumarzouk OM, Monga M, Kata SG, Traxer O, Somani BK. Flexible ureteroscopy and laser lithotripsy for stones >2 cm: a systematic review and meta-analysis. J Endourol. 2012 Oct;26(10):1257-63. doi: 10.1089/end.2012.0217. Epub 2012 Jul 30. PMID 22642568
- [Result] Wong KA, Sahai A, Patel A, Thomas K, Bultitude M, Glass J. Is percutaneous nephrolithotomy in solitary kidneys safe? Urology. 2013 Nov;82(5):1013-6. doi: 10.1016/j.urology.2013.06.034. Epub 2013 Aug 16. PMID 23958507
- [Result] De S, Autorino R, Kim FJ, Zargar H, Laydner H, Balsamo R, Torricelli FC, Di Palma C, Molina WR, Monga M, De Sio M. Percutaneous nephrolithotomy versus retrograde intrarenal surgery: a systematic review and meta-analysis. Eur Urol. 2015 Jan;67(1):125-137. doi: 10.1016/j.eururo.2014.07.003. Epub 2014 Jul 23. PMID 25064687
- [Result] Bas O, Bakirtas H, Sener NC, Ozturk U, Tuygun C, Goktug HN, Imamoglu MA. Comparison of shock wave lithotripsy, flexible ureterorenoscopy and percutaneous nephrolithotripsy on moderate size renal pelvis stones. Urolithiasis. 2014 Apr;42(2):115-20. doi: 10.1007/s00240-013-0615-2. Epub 2013 Oct 27. PMID 24162954
- [Result] Resorlu B, Unsal A, Ziypak T, Diri A, Atis G, Guven S, Sancaktutar AA, Tepeler A, Bozkurt OF, Oztuna D. Comparison of retrograde intrarenal surgery, shockwave lithotripsy, and percutaneous nephrolithotomy for treatment of medium-sized radiolucent renal stones. World J Urol. 2013 Dec;31(6):1581-6. doi: 10.1007/s00345-012-0991-1. Epub 2012 Nov 22. PMID 23179732
- [Result] Ozturk U, Sener NC, Goktug HN, Nalbant I, Gucuk A, Imamoglu MA. Comparison of percutaneous nephrolithotomy, shock wave lithotripsy, and retrograde intrarenal surgery for lower pole renal calculi 10-20 mm. Urol Int. 2013;91(3):345-9. doi: 10.1159/000351136. Epub 2013 Jun 28. PMID 23816573